CLINICAL TRIAL: NCT01877551
Title: Tauroursodeoxycholic Acid for Protease-inhibitor Associated Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201306105; R01DK096982 (NIH)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: HIV Related Insulin Resistance; Protease Inhibitor Related Insulin Resistance; Endoplasmic Reticulum Stress
Keywords: HIV; Protease inhibitor; insulin resistance; Tauroursodeoxycholic acid
MeSH Terms: conditions — Insulin Resistance | interventions — ursodoxicoltaurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tauroursodeoxycholic acid (Active Comparator): This group will receive 1.75 grams per day of tauroursodeoxycholic acid given once daily for 30 days.
  Interventions: Drug: Tauroursodeoxycholic acid
- placebo (Placebo Comparator): This group will receive a placebo tablet that is identical to the treatment group except that it does not contain tauroursodeoxycholic acid. The pills will be taken once daily for 30 days.
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Drug: Tauroursodeoxycholic acid — The intervention group will receive 1.75 grams of tauroursodeoxycholic acid daily for 30 days.
  Other Names: taurolite; tudcabil
  Arms: tauroursodeoxycholic acid
Other: Placebo tablet — The placebo group will receive a placebo tablet that is identical to the treatment group except that it does not contain tauroursodeoxycholic acid. The pills will be taken once daily for 30 days.
  Arms: placebo

SUMMARY:
Rates of cardiovascular disease and diabetes are more than 2-fold greater in HIV infected people than the general population. Protease inhibitor booster antiretroviral therapy (PI-ART) which is used by ~50% of HIV infected people in the USA is an established risk factor for diabetes. Tauroursodeoxycholic acid (TUDCA), a naturally occurring bile salt, improves insulin sensitivity in HIV uninfected subjects, although the mechanisms for these benefits are unclear. This study will explore the hypothesis that TUDCA will improve insulin action in people with HIV who are receiving PI-ART. Further, this project will clarify the molecular mechanisms responsible for these improvements potentially benefiting society, irrespective of HIV status.

DETAILED DESCRIPTION:
The purpose of this study is to determine if, and through which mechanisms, tauroursodeoxycholic acid improves insulin sensitivity in subjects with protease-inhibitor associated insulin resistance.

The investigators will perform body composition analysis by using a DEXA machine, liver fat measurement by using an MRI, and hyperinsulinemic euglycemic clamp procedures in 48 HIV infected, insulin-resistant/prediabetic subjects before and after 30 days of treatment with tauroursodeoxycholic acid or matching placebo. Biopsies of adipose tissue and skeletal muscle will be taken during fasting conditions and during insulin infusion, before and after treatment to measure markers of endoplasmic reticulum stress and thyroid hormone deiodinase.

Outcome measures:

The primary outcome measures will be change in glucose clearance during insulin infusion, change in markers of endoplasmic reticulum stress and change in content of D2 in muscle.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* receiving protease inhibitor containing antiretroviral therapy for >6 months
* Undetectable viral load
* insulin resistant

  1. impaired fasting glucose (fasting blood glucose>100mg/dl)
  2. impaired glucose tolerance (blood glucose >140mg/dl at 2 hours during oral glucose tolerance testing).
* abstained from medications that affect glucose (e.g. prednisone, growth hormone)
* stable medications for >3 months

Exclusion Criteria:

* weight loss of >5% of body weight in prior 6 months
* active gastrointestinal disease (gallstones, pancreatitis, hepatitis, diarrhea)
* use of anti-diabetic medications
* cardiovascular disease (uncontrolled hypertension, heart attack, heart failure, prior endocarditis)
* history of or active substance abuse
* blood clotting disorder or taking medications that affect blood clotting (e.g. coumadin, warfarin)
* pregnant, planning to become pregnant or lactating
* unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic N. Reeds, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Kars M, Yang L, Gregor MF, Mohammed BS, Pietka TA, Finck BN, Patterson BW, Horton JD, Mittendorfer B, Hotamisligil GS, Klein S. Tauroursodeoxycholic Acid may improve liver and muscle but not adipose tissue insulin sensitivity in obese men and women. Diabetes. 2010 Aug;59(8):1899-905. doi: 10.2337/db10-0308. Epub 2010 Jun 3. PMID 20522594
- See also: Washington University AIDS Clinical Trials Unit — http://actu.im.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tauroursodeoxycholic Acid | Placebo
Started | 13 | 14
Completed | 13 | 13
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tauroursodeoxycholic Acid | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants] — Population: one subject in the control group developed influenza during the study and was excluded from final analysis
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 13 | 14 | 27
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 51 (10) | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Glucose Uptake
Description: We will examine the ability of insulin to cause muscle to take up insulin. Each subject will receive intravenous insulin for 6 hours to see how much sugar needs to be given intravenously to keep the blood sugar normal, a measure called glucose uptake. We will compare glucose uptake measured as the amount of 20% dextrose that is needed to keep the blood sugar at ~100mg/dl during insulin infusion before and after 30 days of treatment with drug or placebo.
Time Frame: Glucose uptake is measured at baseline and 30 days after study intervention
Measure: Mean (Standard Error); unit: change in glucose infusion rate (ml/hr)
Arm/Group | Tauroursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 13 | 13
change in glucose infusion rate (ml/hr) | 0 (11) | 8 (7)

2. Secondary Outcome: Body Composition
Description: We will measure how much fat is present in each subject before and after treatment with TUDCA or placebo.
Time Frame: Pre-Treatment and Post 30 day-Treatment
Measure: Mean (Standard Error); unit: percentage of body fat
Arm/Group | Tauroursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 9 | 7
percentage of body fat
  Pre | 35.7 (2.3) | 32.6 (2.8)
  Post | 35.7 (2.3) | 31.7 (2.8)

3. Secondary Outcome: Liver Fat
Description: We will use MRI to measure the relative (%) amount of fat in each subject's liver before and after 30 days of treatment. This will allow us to determine if the drug reduces liver fat. This is calculated by subtracting the amount of fat in the liver at the beginning of the study from the amount of fat in the liver after 30 days of treatment. Subjects who have claustrophobia or are unable to undergo MRI will not have this measure performed. Due to these reasons liver MRS was only performed in 10 patients in the tauroursodeoxycholic acid group and 9 subjects in the placebo group
Time Frame: Pre-Treatment and Post 30 day-Treatment
Measure: Mean (Standard Error); unit: Change in Percent liver fat
Arm/Group | Tauroursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 10 | 9
Change in Percent liver fat | -0.3 (0.2) | 1.2 (0.6)

4. Secondary Outcome: Liver Function Tests
Description: We will measure liver function tests before and after the study drug to ensure that no abnormalities in liver function occurs with the drug.
Time Frame: Pre-Treatment and Post 30 day-Treatment
Measure: Mean (Standard Error); unit: ALT (IU/ml)
Arm/Group | Tauroursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 13 | 13
ALT (IU/ml)
  ALT-PRE | 25 (4) | 21 (2)
  ALT-Post | 19 (3) | 23 (4)

ADVERSE EVENTS:
Time Frame: Adverse event data were taken over a 6 week period after initiation of drug or placebo
Description: Subjects were followed for 6 weeks
Arm/Group | Tauroursodeoxycholic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 1/13 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tauroursodeoxycholic Acid (N=13) | Placebo (N=14)
influenza (Infections and infestations) | 1 (1) | 0 (0) — patient contracted influenza during study

LIMITATIONS AND CAVEATS:
We were unable to recruit our targeted enrollment reducing the power of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT01877551/Prot_SAP_000.pdf